CLINICAL TRIAL: NCT05175417
Title: Visualization of Neural Targets With 3T MRI
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Andres M. Lozano, University Professor, University Health Network, Toronto
Other Study IDs: 21-6105
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Neuro-Degenerative Disease
Keywords: MRI sequence parameters

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients being considered for functional neurosurgical procedures, such as deep brain stimulation (DBS), radiofrequency ablation (RFA), gamma knife radiosurgery (GKR), or magnetic resonance-guided focused ultrasound (MRgFUS).
  Interventions: Other: MRI
- Control: Healthy control volunteers.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — 3 tesla (T) MRI to provide higher resolution and quality brain images.

SUMMARY:
Functional neurosurgery is dedicated to modulating aberrant neural circuits associated with a wide range of neurological conditions. Recently, technological advances in MRI have permitted marked improvements in the direct visualization of neural targets, which is necessary for the accurate targeting in functional neurosurgery procedures.

This research study focuses on imaging patient brains before their scheduled procedures by using a 3 tesla (T) MRI to provide higher resolution and quality brain images. The reason for this study is to assess the image quality using different MRI sequences or settings to improve the image resolution of the most common functional neurosurgery targets (e.g., subthalamic nucleus, globus pallidus, and thalamus) and compare the image quality of the brains in patients with healthy controls. Performing a preoperative MRI is standard-of-care for patients indicated for deep brain stimulation (DBS), gamma knife radiosurgery (GKRS), radiofrequency ablation (RFA), magnetic resonance-guided focused ultrasound (MRgFUS). MRI sequence parameters shown to improve the image quality of different neural structures in a recent literature review (Boutet et al. 2021) will be reproduced on the 3T MRI at Toronto Western Hospital.

DETAILED DESCRIPTION:
This is an exploratory prospective experimental study that will assess the ability of different MRI sequences to visualize common functional neurosurgical targets. Some neural structures (i.e., STN) are sometimes not visualized as well, particularly in older patients, when compared to healthy controls. The findings from this study should help in identifying the advanced sequences for direct visualization of these targets, that could then be used for improved preoperative planning of functional neurosurgical procedures.

Several advanced MRI sequences will be conducted when imaging patients or healthy participant. All advanced sequences have previously been published in the literature as viable, safe preoperative planning sequences for functional neurosurgical treatments at other centres. All MRI scans in this study will be acquired at the Toronto Western Hospital (TWH). For example, structural scans using sequences that can null or not receive signals from fluids in the brain and reduce geometric distortion (i.e., fluid attenuated inversion recovery (FLAIR)), null white matter signals (i.e., fast gray matter acquisition T1 inversion recovery (FGATIR)), and enhance the visualization of iron concentrated neural structures (i.e., quantitative susceptibility mapping (QSM)) will be performed. These advanced sequences will be compared to conventional structural MRI sequences (i.e., T1-weighted (T1W) or T2-weighted (T2W)) that are typically used for anatomical purposes and direct visualization of neural structures.

Ultimately, results from this study should enhance quality of care, clinical benefits, and data quality.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years of age.
* Preparing to undergo a functional neurosurgical intervention (e.g., DBS, RFA, GKR or MRgFUS) at TWH (not applicable for healthy volunteers).
* Participants must be able to understand the purpose of this research and must sign the informed consent form.
* Participants must understand that the role of this research is to enhance our understanding of brain functioning and that he/she will not directly or indirectly benefit from the study.

Exclusion Criteria:

* Contraindication for an MRI (e.g., implanted cardiac device, metal in eyes, aneurysm clip, etc.).
* Participants who have serious cognitive or psychological impairments and cannot give informed consent.
* Participants who are unable to communicate effectively or efficiently (e.g., patients suffering from speech deficits (dysarthria, aphasia) or are non-English speaking).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients indicated for deep brain stimulation (DBS), radiofrequency ablation (RFA), gamma knife radiosurgery (GKR), or magnetic resonance-guided focused ultrasound (MRgFUS).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-01-29 (Actual); Primary Completion 2024-08-29 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative image quality metrics | ≤ 1 week before surgery
  Two quantitative image quality metrics commonly used are contrast-to-noise ratio (CNR) and signal-to-noise ratio (SNR). CNR (i.e., the ratio of the contrast between the signal in a given region and the background) is a measure of the contrast between the tissue of interest and the neighboring tissue. Similarly, SNR is a measure of the average image signal in a given region to the neighboring tissue or the noise around the region of interest.
Qualitative image quality metrics | ≤ 1 week before surgery
  Qualitative image quality metrics will assess the image quality and clinical acceptability of each scan in a randomized order. Each scan will be scored using a 5-point Likert scale by expert raters. An overall average score will be calculated for each MRI sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Andres M Lozano, MD/PhD, Principal Investigator — University Health Network, Toronto, ON
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boutet A, Loh A, Chow CT, Taha A, Elias GJB, Neudorfer C, Germann J, Paff M, Zrinzo L, Fasano A, Kalia SK, Steele CJ, Mikulis D, Kucharczyk W, Lozano AM. A literature review of magnetic resonance imaging sequence advancements in visualizing functional neurosurgery targets. J Neurosurg. 2021 Mar 26;135(5):1445-1458. doi: 10.3171/2020.8.JNS201125. Print 2021 Nov 1. PMID 33770759
- See also: A literature review of magnetic resonance imaging sequence advancements in visualizing functional neurosurgery targets — http://pubmed.ncbi.nlm.nih.gov/33770759/